CLINICAL TRIAL: NCT02281175
Title: The Effectiveness of a Novel Psychosocial Intervention "Programme d'Aide au Succès du Sevrage " (PASSE-65+) Designed to Help Older Benzodiazepine Users to Gradually Wean Their Medication
Brief Title: How to Ease the Withdrawal of Tranquilizers Among Older Consumers?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre de Recherche de l'Institut Universitaire de Geriatrie de Montreal (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Universite du Quebec en Outaouais (Other); Université de Montréal (Other); Université de Sherbrooke (Other); Laval University (Other)
Responsible Party: Principal Investigator, Dr Sébastien Grenier, Research Associate Professor, Centre de Recherche de l'Institut Universitaire de Geriatrie de Montreal
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CRIUGM-003
Record Dates: First submitted 2014-10-22; First posted 2014-11-03 (Estimated); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Drug Dependence
Keywords: Benzodiazepine withdrawal; PASSE-65+ program; Psychosocial (non-pharmacological) intervention; Cognitive-Behavioral Therapy (CBT); Older adults
MeSH Terms: conditions — Substance-Related Disorders | interventions — Psychosocial Intervention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- No contact intervention (No Intervention): Informative document that proposes a 12-week self-withdrawal grid
- a weekly physician intervention (Active Comparator): Informative document + 12 meetings (once a week; 30 minutes) with a physician who will supervise the gradual withdrawal
  Interventions: Behavioral: a weekly physician intervention
- psychosocial intervention (Experimental): Informative document + 12 meetings (once a week; 30 minutes) with a physician who will supervise the gradual withdrawal + psychosocial intervention (PASSE-65+ program: 12 sessions over 16 weeks)
  Interventions: Behavioral: Psychosocial intervention

INTERVENTIONS:
Behavioral: Psychosocial intervention — Based on a cognitive-behavioral approach, the psychosocial intervention (PASSE-65+) is specifically designed to help older BZD users to better manage their withdrawal symptoms, to stop their medication, and to improve their general psychological well-being
  Arms: psychosocial intervention
Behavioral: a weekly physician intervention — Informative document + 12 meetings (once a week; 30 minutes) with a physician who will supervise the gradual withdrawal
  Arms: a weekly physician intervention

SUMMARY:
Benzodiazepines (BZD) are widely used to treat anxiety, insomnia, and depression. These drugs can have very serious side effects if they are taken over a long period of time. In addition to stability, memory, concentration, vigilance, and attention impairments, long-term use of BZD is also associated with an increased in hypertension incidence, urinary incontinence, coronary artery disease, and renal complications. There are growing evidences that long-term BZD use causes physical and psychological dependence as evidenced by the withdrawal syndrome.

The recommended strategy by physicians to facilitate the withdrawal of BZD is to gradually reduce the medication, either by replacing the BZD by another with a longer half-life, or by the gradual dose reduction. Unfortunately, the success of such a procedure is low as up to 80% of people who try to quit, relapse due to the intolerance of withdrawal symptoms. Therefore, it is important to find new strategies to overcome the withdrawal difficulties.

The aim of this study is to test the effectiveness of a novel psychosocial intervention called PASSE-65+ to facilitate the benzodiazepine withdrawal in the older users, thus providing a new therapeutic tool to physician.

DETAILED DESCRIPTION:
Benzodiazepines (BZD) represent the most frequently consumed drugs by the elderly persons in Canada. Indeed, there is 7.5 times more BZD users in older people (65 years and over) than in adults (18-64 years). Importantly, more than 50% of seniors who received a prescription of BZD do not display any severe psychiatric symptoms and are physically in good health.

Results from a survey including 2811 community-dwelling older adults (65 years and over) showed that 32% of the respondents consumed BZD for an average of 205 days and 60% of them had at least received one potentially inappropriate prescription during this period (e.g. a prescription of a BZD with a long half-life or a prescription of 2 BZD for more than 6 consecutive weeks, etc.). Another study showed that 45% of new BZD users take these drugs for more than 30 days. It should be noted that the definition of a long-term BZD use varies from three to four months of consumption, which corresponds to the average period used by almost all seniors.

Long-term use of BZD by older people is a complex phenomenon that can be explained by several personal, psychological, and social factors interacting with each other. Systemic model of BZD consumption in late-life implies the following five elements which contribute to initiate and maintain BZD taking: 1) history (i.e. autonomy loss, stress, disease apparition, etc.); 2) the prescription process; 3) personal dispositions (i.e. sexe, age, education, loneliness, etc.); 4) sociocultural factors (i.e. positive attitude of their family or their physician toward BZD use); and 5) cognitive strategies (e.g. trivialization of concerns about the drugs, etc.).

To the researcher's knowledge, very few randomized controlled clinical trials have tested the effectiveness of non-pharmacological interventions in patients with a mean age of 60 years and older. Data from these studies showed that brief intervention (e.g. receiving either an informative leaflet on BZD withdrawal during a meeting with the doctor or an informative letter by post mail) or psychological interventions (including cognitive behavioral therapy or CBT) are most likely more effective than the standard care and in some cases, to the gradual dose reduction (GDR) supervised by a physician. However, only 10% (brief intervention) to 85% (cognitive behavioral therapy designed to treat insomnia) of participants completely stopped BZD use at the end of treatment. Furthermore, Parr and colleagues indicate that the complete stop of BZD consumption remains difficult and still a big challenge to patients, clinicians and researchers.

Nevertheless, one of the limitations of these studies is the large variation of age of their participants (ranging from 18 to 85 years, despite a mean age of over 60 years), thus restricting the generalization of the findings to older patients. Moreover, these results derive from efficacy studies (vs effectiveness studies) designed to improve internal validity at the expense of external validity. Although these results demonstrate the potential efficacy (vs effectiveness) of non-pharmacological treatments to facilitate BZD withdrawal, very few elderly users receive such interventions due to lack of resources, expertise and time or simply due to their expensive implementation cost. Finally, to the investigator's knowledge, no psychosocial intervention based on cognitive-behavioral therapy (CBT) and including other specific personal, psychological, and social components associated to aging, and targeting older people with different psychological problems (i.e. not only insomnia but also anxiety or depression) has been tested. Therefore, the researcher hypothesized that the "Programme d'Aide au Succès du SEvrage (PASSE-65+)" could be more suitable and effective to help older people in their BZD withdrawal management.

In order to answer the investigator's hypothesis, long-term older users of BZD will first receive a clinical assessment to determine whether they meet the research criteria. The participants (n=75) will then be randomly allocated to one of the following three groups: one group will receive an informative document (describing the steps for a gradual self-weaning), a second will receive the same informative document and will have a 30 minutes meeting with a physician once a week, and the third group will receive the informative document, will meet a physician once a week and will receive a psychosocial intervention (PASSE-65+).

It is noteworthy that the psychosocial intervention will also be offered to the first 2 groups at the end of the study.

The research study will be conducted during a 12 week-period for the first 2 groups. For the third group, the intervention will be offered on 12 sessions during a 16 week-period.

All groups will undergo three additional assessments (2 to 14 days, 3 months and 12 months) following end of interventions. These last assessments aim to measure the rate of relapse, withdrawal symptoms, intensity of anxious and depressive symptoms, and the sleep quality of participants.

Finally, 15 participants will be randomly chosen and divided into 3 groups (n=5): One group will be constituted by BZD users who completely stopped taking their drug, the second one with BZD users who diminished their consumption and the third one with participants who relapsed or dropped out. All participants from these groups will be interviewed at home to collect their opinion about the PASSE-65+ program.

ELIGIBILITY:
Inclusion Criteria:

* Be aged 65 years and older;
* To consume benzodiazepine for at least two years (even if consumption is not continuous);
* Want to quit benzodiazepine use.

Exclusion Criteria:

* Living a difficult situation that requires specific interventions (e.g. bereavement or death, a recent breakup or suicidal thoughts);
* Alcohol or illicit drugs addiction (other than benzodiazepine);
* BZD use for medical reasons (e.g. epilepsy);
* Be unable to complete the questionnaires or to attend meetings for any reason (e.g. Loss of vision, severe arthritis, cognitive impairment, etc.).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 114 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Change in consumed BZD (diazepam equivalent) dose | 1 month before the beginning of the intervention and 2-14 days, 3 months and 12 months after the end of intervention (a total of four assessments)
  Comparison between the average dose of BZD (diazepam equivalent) consumed during the month preceding the beginning of intervention and the one consumed between 2-14 days , 3 months and 12 months after the end of intervention.

SECONDARY OUTCOMES:
Assessment of withdrawal symptoms | 1 month before the beginning of the intervention and 2-14 days, 3 months and 12 months after the end of intervention (a total of four assessments)
  Benzodiazepine Withdrawal Symptom Questionnaire (BWSQ)
Evaluation of self-competence OU self-confidence towards change in benzodiazepine use | 1 month before the beginning of the intervention and 2-14 days, 3 months and 12 months after the end of intervention (a total of four assessments)
  Perceived Competence Scale (PCS)
Estimation of attitudes towards benzodiazepine consommation | 1 month before the beginning of the intervention and 2-14 days, 3 months and 12 months after the end of intervention (a total of four assessments)
  Attitudes Towards Tranquilizer Use Questionnaire (ATTUQ)
Symptoms of anxiety OU worry assessment | 1 month before the beginning of the intervention and 2-14 days, 3 months and 12 months after the end of intervention (a total of four assessments)
  Penn State Worry Questionnaire (PSWQ)
Measurement of depression symptoms | 1 month before the beginning of the intervention and 2-14 days, 3 months and 12 months after the end of intervention (a total of four assessments)
  Beck Depression Inventory-II (BDI-II)
Assessment of sleep quality | 1 month before the beginning of the intervention and 2-14 days, 3 months and 12 months after the end of intervention (a total of four assessments)
  Pittsburgh Sleep Quality Index (PSQI)

OTHER OUTCOMES:
Economic cost analysis | 12 months before the beginning of the intervention, during the intervention and 12 months after the end of intervention
Cost analysis related to the health system and to the patient | 12 months before the beginning of the intervention, during the intervention period and 12 months after the end of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien Grenier, Ph.D., Principal Investigator — Centre de Recherche de l'Institut Universitaire de Geriatrie de Montreal
Locations (1):
- Centre de Recherche de l'Institut Universitaire de Geriatrie de Montreal, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Allary A, Proulx-Tremblay V, Belanger C, Hudon C, Marchand A, O'Connor K, Perodeau G, Roberge P, Tannenbaum C, Vasiliadis HM, Desrosiers C, Cruz-Santiago D, Grenier S. Psychological predictors of benzodiazepine discontinuation among older adults: Results from the PASSE 60. Addict Behav. 2020 Mar;102:106195. doi: 10.1016/j.addbeh.2019.106195. Epub 2019 Oct 31. PMID 31838367
- [Derived] Proulx-Tremblay V, Allary A, Payette MC, Benyebdri F, Boudreau MM, Bernard C, Leveille V, Desrosiers C, Cruz-Santiago D, Gagne MH, Bertrand JA, Grenier S. Social support and sleep quality in older benzodiazepine users. Aging Ment Health. 2020 Sep;24(9):1437-1443. doi: 10.1080/13607863.2019.1594167. Epub 2019 Apr 12. PMID 30977682
- See also: Lab website (in french only) — http://www.laboleader.ca